CLINICAL TRIAL: NCT06938321
Title: An Open Label, Multicenter, Phase Ib/II Clinical Study of AK130 in Combination With AK112 for the Treatment of Advanced Biliary Tract Cancer
Brief Title: A Study of AK130 in Combination With AK112 for the Treatment of Advanced Biliary Tract Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK130-201
Record Dates: First submitted 2025-03-10; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK112 in combination with AK130 (Experimental)
  Interventions: Drug: AK112; Drug: AK130
- AK112 (Experimental)
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — Following a predefined dose and date.
Drug: AK130 — Following a predefined dose and date.
  Arms: AK112 in combination with AK130

SUMMARY:
There're 2 parts in this interventional study:

1. The goal of phase Ib trial is to evaluate the safety and tolerability of AK130 in combination with AK112 therapy for the purpose of observing the incidence of dose limit toxicity (DLT) as well as the confirmation of maximum tolerable dose (MTD) in the treatment of advanced biliary tract cancer (BTC), so as to determine the recommended phase 2 dose (RP2D) in the second part of the trial.
2. The goal of phase II trial is to evaluate the safety and efficacy of AK112 in combination with AK130 therapy or monotherapy in the treatment of advanced BTC.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent.
2. Have a life expectancy of at least 3 months.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Subjects with histologically and/or cytologically confirmed advanced or metastatic biliary tract malignancies (including only intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder carcinoma; excluding ampullary carcinoma), who have experienced treatment failure following prior first-line systemic therapy.
5. According to RECIST v1.1, there is at least one untreatable measurable lesion, or a measurable lesion with clear imaging progression after local treatment, suitable for repeated and accurate measurement.
6. Has adequate organ function.
7. All subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.
8. Able to to comply with all requirements of study participation (including all study procedures).

Exclusion Criteria:

1. Except for BTC, the subjects had other malignant tumors within the 3 years prior to enrollment. Subjects with other malignant tumors that have been cured through local treatment are not excluded, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical or breast cancer in situ.
2. There is central nervous system (CNS) metastasis, spinal cord compression, or meningeal metastasis.
3. There are pleural effusion, pericardial effusion, or ascites with clinical symptoms or requiring repeated drainage.
4. Prior administration of any immunotherapy targeting immune mechanisms other than PD-1/PD-L1 inhibitors.
5. There is a history of non infectious pneumonia that requires systemic glucocorticoid treatment.
6. History of severe bleeding tendency or coagulation dysfunction.
7. Previous history of myocarditis, cardiomyopathy, and malignant arrhythmia.
8. Any arterial or severe venous thromboembolism events, transient ischemic attacks, cerebrovascular accidents, hypertensive crises, or hypertensive encephalopathy occurred within 6 months prior to the first administration of medication.
9. Pregnant or lactating female subject.
10. Any prior or concurrent disease, treatment, or laboratory test abnormality that may confuse study results, affect subjects' full participation in the study, or may not be in their best interest to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities (DLTs) | During the first three weeks.
  DLTs will be assessed during the first three weeks of treatment. DLTs are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the DLT observation period.
Number of subjects with adverse events (AEs) | From the time of informed consent signed through 30 days after the last dose of study drug or starting new anti-cancer therapy.
  AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.
Objective Response Rate (ORR) (Phase II) | Through study completion, an average of 2 years.
  ORR is defined as the proportion of subjects with BOR response of CR or PR (based on RECIST Version 1.1).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (Phase Ib) | Through study completion, an average of 2 years.
  ORR is defined as the proportion of subjects with BOR response of CR or PR (based on RECIST Version 1.1).
Disease control rate (DCR) | Through study completion, an average of 2 years
  DCR is defined as the proportion of subjects with response of CR, PR and SD (based on RECIST Version 1.1).
Duration of Response (DoR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The time from first documented evidence of CR or PR until time of first documented disease progression.
Time to response (TTR) | From date of randomization until the date of first documented response, assessed up to 24 months
  Time between date of start of treatment until first documented response (CR or PR).
Progression Free Survival (PFS) | Through study completion, an average of 2 years.
  PFS is defined as the interval between first dose and the earliest date of disease progression or death due to any cause.
Overall survival (OS) | Through study completion, an average of 2 years.
  OS is defined as the time from first dose until death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No